CLINICAL TRIAL: NCT03108326
Title: Real World Effectiveness of Ustekinumab in Induction and Maintenance Therapy for Crohn´s Disease in Conjunction With Long-term Outcome
Brief Title: Real World Effectiveness of Ustekinumab in Induction and Maintenance Therapy for Crohn´s Disease
Acronym: RUN-CD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ced Service GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: bio101
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab; Infliximab; vedolizumab; Adalimumab; CT-P13

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (6):
- Group 1a: CD-patients (age at enrollment: 18-80 years) receiving a newly introduced Ustekinumab therapy (n=150). A prior therapy with biologics is not allowed.
- Group 1b: CD-patients (age at enrollment: 18-80 years) receiving a newly introduced Ustekinumab therapy (n=150). A prior therapy with 1 biologics is allowed
- Group 2: CD-patients (age at enrollment: 18-80 years) receiving a newly introduced Ustekinumab therapy (n=150). A prior therapy with ≥2 biologic is allowed.
  Interventions: Biological: Stelara, Remicade, Entyvio, Humira, Remsima, Flixabi, Inflectra
- Group 3a: CD-patients (age at enrollment: 18-80 years) receiving a newly introduced biologics therapy other than Ustekinumab (n=150). A prior therapy with biologic is not allowed.
- Group 3b: CD-patients (age at enrollment: 18-80 years) receiving a newly introduced biologics therapy other than Ustekinumab (n=150). A prior therapy with 1 biologic is allowed.
- Group 4: CD-patients (age at enrollment: 18-80 years) receiving a newly introduced biologics therapy other than Ustekinumab (n=150). A prior therapy with ≥2 biologics is allowed.
  Interventions: Biological: Stelara, Remicade, Entyvio, Humira, Remsima, Flixabi, Inflectra

INTERVENTIONS:
Biological: Stelara, Remicade, Entyvio, Humira, Remsima, Flixabi, Inflectra — The data of Crohn´s Disease (CD)-patients on Ustekinumab will be compared in an explorative analysis with CD-patients on other Biologics.
  Groups: Group 2; Group 4

SUMMARY:
"RUN-CD" is an investigator initiated "Non interventional Trial" on biologics in Crohn´s Disease (CD) patients in Germany with a prospective documentation of effectiveness in induction and maintenance therapy of biologics, especially of Ustekinumab, with a special interest on predictors of long-term responses and favorable disease outcome and documentation of severe side effects caused by the therapy with biologics.

DETAILED DESCRIPTION:
The effectiveness and safety of induction and maintenance therapy of Ustekinumab and other biologics will be assessed in different relevant subgroups of Crohn's Disease patients. To this end, different confounders have to be considered. Patients followed-up for several years will likely receive changing treatments. These changes have to be taken into account. Furthermore, the decision to prescribe, to stop or to continue a treatment depends on the availability of treatment options and experiences with these alternatives:

1. Confounding by indication will be taken into account
2. Patient characteristics which likely influence the risk of developing a particular endpoint will be taken into account
3. The possible influence of co-medication will be considered
4. Changing risks over time will be considered
5. Power considerations needs to be conducted prior to the comparison of incidence rates
6. Appropriate statistical methods will be applied to deal with these challenges

The principles described above will be followed in a similar manner for the analysis of effectiveness and safety endpoints. An appropriate power analysis will be performed before each sub-analysis.

ELIGIBILITY:
Inclusion Criteria:

CD-patients aged 18-80 years at enrollment written informed consent is given

Exclusion Criteria:

planned surgical intervention malignant disease in history lack of adequate documentation possibilities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Crohn´s Disease (CD)-patients will be prospectively documented in the post-marketing observational investigator initiated study (RUN-CD). The diagnosis is made in accordance with current DGVS/ECCO CD-guidelines.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of induction therapy in CD-patients treated with Ustekinumab. | Week 0 till 16
  clinical remission HBI ≤ 4 at week 16

SECONDARY OUTCOMES:
Effectiveness of induction therapy at week 8 in CD-patients treated with Ustekinumab vs. anti-TNF/Vedolizumab. | Week 0 till 8
  clinical remission HBI ≤ 4 at week 8
Effectiveness of maintenance therapy up to 3 years in CD-patients treated with Ustekinumab vs. anti-TNF/Vedolizumab. | Week 0 till year 3
  clinical remission HBI ≤ 4 at year 3
Effectiveness of Ustekinumab in different subpopulations | Week 0 till year 3
  e.g. based on prior biologics therapy or clinical parameters/phenotype at baseline in comparison with the other biologics-group.
  or clinical parameters/phenotype at baseline in comparison with the other biologics-group.
Measurement of disease activity with HBI | Week 0 till year 3
  HBI= Harvey-Bradshaw-Index (e.g. steroids), co-morbidities and adverse events.
Measurement of Quality of Life with EQ-5D questionnaire | Week 0 till year 3
  EQ-5D™ is a standardised instrument for use as a measure of health outcome
Measurement of disease activity with CDAI | Week 0 till week 16
  CDAI = Crohn's Disease Activity Index

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterologische Gemeinschaftspraxis Minden, Minden, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided